CLINICAL TRIAL: NCT07165743
Title: Negative Predictive Value of Rapid Emptying of the Fetal Bladder (≤40 Min and Post-void ≤2 mm) on Major Chromosome Aneuploidies at 11-14 Gestational Weeks: A Prospective Diagnostic Accuracy Study
Brief Title: Evaluation of Fetal Bladder Emptying During the 11-14 Weeks' Ultrasound Examination as a Negative Predictive Marker for Chromosomal Abnormalities
Status: Active, not recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Can Bilginer, Fellow at Perinatology department, Haseki Training and Research Hospital
Other Study IDs: HasekiTRH 27.08.2025 155-2025
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chromosomal Aneuploidies (e.g., Trisomy 21, Trisomy 18, Trisomy 13); Prenatal Screening Accuracy
Keywords: First-trimester screening Chromosomal abnormalities Prenatal diagnosis Ultrasound Negative predictive value (NPV) Fetal bladder
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 270 Months

GROUPS / COHORTS (2):
- Pregnancies in which the fetal bladder empties completely within ≤ 40 minutes
  Interventions: Diagnostic Test: 40-Minute Real-Time First-Trimester Ultrasonography
- Pregnancies in which the bladder does not meet the rapid-emptying criteria
  Interventions: Diagnostic Test: 40-Minute Real-Time First-Trimester Ultrasonography

INTERVENTIONS:
Diagnostic Test: 40-Minute Real-Time First-Trimester Ultrasonography — A one-time midsagittal ultrasound performed between 11 +0 and 14 +0 weeks. Bladder emptying time and post-void longitudinal bladder diameter are recorded. No invasive procedures are performed.

SUMMARY:
Template-Based Brief Summary (Sağlık Profesyonelleri İçin)

Study Title:

The Negative Predictive Value of First-Trimester Fetal Bladder "Rapid Emptying" (≤40 minutes and post-void ≤2 mm) for Major Chromosomal Aneuploidies: A Prospective Diagnostic Accuracy Study.

Purpose:

To evaluate whether the dynamic phenotype of rapid bladder emptying at 11-14 weeks reduces the likelihood of major chromosomal abnormalities (particularly Trisomy 21) compared to fetuses without this phenotype.

Design:

Single-center, prospective observational cohort.

Population:

270 singleton pregnancies between 11+0 and 14+0 weeks.

Procedures:

Real-time sagittal ultrasound observation for 40 minutes.

Documentation of bladder emptying time and post-void longitudinal bladder diameter.

Concurrent measurement of CRL, NT, ductus venosus waveform.

Gold standard confirmation with cfDNA or invasive karyotyping in high-risk cases.

Primary Endpoint:

Negative predictive value (NPV), ROC-AUC, sensitivity/specificity for aneuploidy detection.

Secondary Endpoints:

Rate of invasive testing, performance in combined models with cfDNA and biophysical markers, Net Reclassification Index.

Duration:

5 months (08/2025 - 01/2026).

Potential Impact:

If validated, the rapid emptying phenotype may serve as a low-risk marker, reduce unnecessary invasive procedures, and refine first-trimester screening algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, viable pregnancy between 11 + 0 and 14 + 0 gestational weeks (GA)
* Maternal age 18 - 45 years at enrollment
* Able to provide written informed consent

Exclusion Criteria:

* Multiple gestation (twins, higher order)
* Major fetal structural anomaly detected at index scan
* Known serious maternal comorbidity (e.g., insulin-dependent diabetes, uncontrolled hypertension, renal or autoimmune disease)
* Participation in another interventional research study during the current pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prospective cohort of 270 consecutive healthy pregnant women with singleton fetuses, attending first-trimester screening (11 - 14 GA) at a tertiary perinatology center in Istanbul, Türkiye.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value (NPV) of Rapid Fetal Bladder Emptying for Detecting Major Chromosomal Aneuploidy | From enrollment at 11 + 0 to 14 + 0 gestational weeks until definitive genetic result or delivery, whichever comes first (≈ 26 weeks).
  Proportion of fetuses with the rapid-emptying phenotype (≤ 40-minute complete emptying + post-void longitudinal bladder diameter ≤ 2 mm) who are subsequently confirmed not to have a major chromosomal aneuploidy (Trisomy 21, 18, or 13) by cfDNA, invasive karyotype, or postnatal testing.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Haseki Training and Research Hospital - Perinatology Department, Istanbul, Istanbul (Sultangazi District), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome analyses-including fetal bladder emptying time, post-void longitudinal bladder diameter, nuchal translucency, ductus venosus waveform, cfDNA results, and karyotype confirmation-will be shared with qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD, çalışma protokolü, SAP ve boş ICF; ana sonuçların hakemli dergide yayımlanmasından itibaren 12 ay içinde erişime açılacak ve 5 yıl süreyle paylaşılabilir olacaktır (yaklaşık Temmuz 2027 - Temmuz 2032).

REFERENCES:
- [Background] Capone V, Persico N, Berrettini A, Decramer S, De Marco EA, De Palma D, Familiari A, Feitz W, Herthelius M, Kazlauskas V, Liebau M, Manzoni G, Maternik M, Mosiello G, Schanstra JP, Vande Walle J, Wuhl E, Ylinen E, Zurowska A, Schaefer F, Montini G. Definition, diagnosis and management of fetal lower urinary tract obstruction: consensus of the ERKNet CAKUT-Obstructive Uropathy Work Group. Nat Rev Urol. 2022 May;19(5):295-303. doi: 10.1038/s41585-022-00563-8. Epub 2022 Feb 8. PMID 35136187
- [Background] Arasaratnam M, Balakrishnar B, Crumbaker M, Turner S, Hayden AJ, Brooks A, Patel MI, Lau H, Woo H, Bariol S, Gurney H. Patterns of care and outcomes of men with germ cell tumors in a high-volume Australian center. Asia Pac J Clin Oncol. 2022 Apr;18(2):e23-e31. doi: 10.1111/ajco.13548. Epub 2021 Jun 21. PMID 34152083
- [Background] Muller K, Kufner K, Prange K, Bengel J. [Screening for Anxiety in People with an Intellectual Disability: German Version of the "Glasgow Anxiety Scale for People with an Intellectual Disability" (GAS-ID)]. Psychiatr Prax. 2019 Jul;46(5):274-280. doi: 10.1055/a-0843-3373. Epub 2019 Mar 19. German. PMID 30891726
- [Background] Zhu R, Lv W, Sun C, Qin C, Zhang D, Long Z. A facile strategy to fabricate high-barrier, water- and oil-repellent paper with carboxymethyl cellulose/collagen fiber/modified polyvinyl alcohol. Carbohydr Polym. 2023 Aug 15;314:120933. doi: 10.1016/j.carbpol.2023.120933. Epub 2023 Apr 20. PMID 37173031
- [Background] Savarese JJ, Tabler NG Jr. Multimodal analgesia as an alternative to the risks of opioid monotherapy in surgical pain management. J Healthc Risk Manag. 2017 Jul;37(1):24-30. doi: 10.1002/jhrm.21262. PMID 28719091
- [Background] Chasserant P, Gosgnach M. Improvement of peri-operative patient management to enable outpatient colectomy. J Visc Surg. 2016 Nov;153(5):333-337. doi: 10.1016/j.jviscsurg.2016.07.006. Epub 2016 Sep 23. PMID 27671006
- [Background] Lesieur E, Barrois M, Bourdon M, Blanc J, Loeuillet L, Delteil C, Torrents J, Bretelle F, Grange G, Tsatsaris V, Anselem O. Megacystis in the first trimester of pregnancy: Prognostic factors and perinatal outcomes. PLoS One. 2021 Sep 7;16(9):e0255890. doi: 10.1371/journal.pone.0255890. eCollection 2021. PMID 34492029